CLINICAL TRIAL: NCT04683926
Title: A Phase 1 Randomized Single Oral Dose Cross-Over Study Investigating Desmetramadol Dose Proportionality And Food Effect In Normal Human Subjects
Brief Title: A Randomized Study Investigating Oral Desmetramadol Dose Proportionality and Food Effect In Normal Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: Celerion (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Omni-Pain-103; R44DA046316 (NIH)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Pain
Keywords: Pharmacokinetics; Food effect
MeSH Terms: conditions — Pain | interventions — O-demethyltramadol

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, balanced, single-dose, four-treatment, four-period, four-sequence (using a Williams' square design) cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Desmetramadol 10 mg, fasted (Experimental): While fasting a single oral dose of 10 mg desmetramadol under.
  Interventions: Drug: Desmetramadol
- Desmetramadol 20 mg, fasted (Experimental): While fasting a single oral dose of 20 mg desmetramadol.
  Interventions: Drug: Desmetramadol
- Desmetramadol 30 mg , fasted (Experimental): While fasting a single oral dose of 30 mg desmetramadol.
  Interventions: Drug: Desmetramadol
- Desmetramadol 30 mg , fed (Experimental): After feeding a single oral dose of 30 mg desmetramadol.
  Interventions: Drug: Desmetramadol

INTERVENTIONS:
Drug: Desmetramadol — Analgesic
  Other Names: Omnitram

SUMMARY:
The purpose of the study is to investigate in healthy human subjects how much desmetramadol (Omnitram) gets in the blood after different oral doses are taken with or without food.

DETAILED DESCRIPTION:
An open-label, randomized, balanced, single-dose, four-treatment, four-period, four-sequence (using a Williams' square design) cross-over study with each dose separated by >3 days. There are 4 sequences (Sequence 1, Sequence 2, Sequence 3, and Sequence 4), and 4 Periods (Period I, Period II, Period III, and Period IV). Sequence 1 order is 30 mg dose with food (Period I); 30 mg dose fasted (Period II), 10 mg dose fasted (Period III), and 20 mg dose fasted (Period IV). Sequence 2 order is 10 mg dose fasted (Period I); 30 mg dose with food (Period II), 20 mg dose fasted (Period III), and 30 mg dose fasted (Period IV). Sequence 3 order is 20 mg dose fasted (Period I); 10 mg dose fasted (Period II), 30 mg dose fasted (Period III), and 30 mg dose with food (Period IV). Sequence 4 order is 30 mg dose fasted (Period I); 20 mg dose fasted (Period II), 30 mg dose with food (Period III), and 10 mg dose fasted (Period IV).

To account for potential dropouts, up to 32 eligible subjects will be randomized to obtain a target sample of 24 subjects with PK responses at each of the four treatment periods (based on our completed phase 1 study in 43 subjects, dropouts are unlikely (~5%); see Section 1.2.2). Before each oral dose, subjects will be fasted overnight for at least 10 hours. Treatment sequences will include the following four unblinded single-dose oral treatments: 1) desmetramadol 1 x 10 mg tablet; 2) desmetramadol 2 x 10 mg tablets; 3) desmetramadol 3 x 10 mg tablets; and 4) desmetramadol 3 x 10 mg tablets following a high-fat, high-calorie breakfast served approximately 30 minutes before dosing and entirely consumed within 20 minutes. All subjects will fast for an additional four hours after desmetramadol administration. The fed treatment should be administered the desmetramadol dose approximately 30 minutes after the start of the meal. Desmetramadol will be administered with approximately 240 ml of water. No water is allowed one hour before and one hour after each desmetramadol administration.

This will be an inpatient study. Subjects will be admitted to the clinical pharmacology unit on Study Day -1, and administered a single oral dose treatment on Study Day 1, Study Day 4, Study Day 7 and Study Day 10. After completing study procedures on Day 11 the subject will be discharged from the facility.

Blood specimens for plasma preparation and PK analysis will be collected at the following times: pre-dose (0 h), and post-dose 0.5, 1.0, 1.5, 2.0, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, and 32 h.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females with vital signs as follows at screening: systolic blood pressure > 90 mm Hg and < 140 mm Hg; diastolic blood pressure > 40 mm Hg and < 90 mm Hg; pulse 40 to 99 beats per minute; respiratory rate 12 to 24 breathes per minute.
2. Age 19 to 55 years.
3. Able and willing to give informed consent
4. Able to comply with all study procedures.
5. If female, must not be of childbearing potential or must agree to use one or more of the following forms of contraception from screening, throughout the study and for 30 days following study drug administration: hormonal (e.g., oral, transdermal, intravaginal, implant or injection for 3 months); double barrier (e.g., condom or diaphragm with spermicide); intrauterine device (IUD) or system (IUS) (for 3 months); vasectomized partner (6 months minimum); or abstinence.

   Screening laboratory results must be within normal range per clinical research unit: serum sodium, potassium, calcium, BUN, creatinine, ALT, AST, total bilirubin, alkaline phosphatase, glucose (random), albumin, total protein, WBC and differential, hemoglobin, and platelets. In addition PT and PTT must be < 1.2 ULN.
6. Electrocardiogram (ECG) without clinically significant abnormalities.

   Urinalysis demonstrating < +1 glucose, and +1 protein.
7. If female, must have a negative pregnancy test at screening
8. Negative urine test for substances of abuse, including opiates, per clinical pharmacology unit standards at screening and clinic check-in.
9. Negative serology tests for HIV, hepatitis B surface antigen, and hepatitis C virus antibody.
10. Weight > 50 Kg and a body mass index (BMI) of 18.0 to 32.0 kg/m (inclusive).
11. Non-smoker of tobacco for a minimum of the past 3 months, and negative urine continine test.

Exclusion Criteria:

1. Oral temperature > 38°C or current illness.
2. History of seizures, epilepsy, or recognized increase risk of seizure (e.g., head trauma, metabolic disorders, alcohol or drug withdrawal).
3. History of cirrhosis or laboratory evidence of liver disease.
4. Having undergone gall bladder removal.
5. Use of alcohol within 24 hours of day -1 until the end of the study; and grapefruit, grapefruit-related citrus fruits (e.g., Seville oranges, pomelos), or grapefruit juice or grapefruit-related juices within 7 days of study drug administration and until the end of the study.
6. History of previous anaphylaxis, severe allergic reaction to tramadol, codeine, or other opioid drugs.
7. Any other unstable acute or chronic disease that could interfere with the evaluation of the safety of the study drug as determined by the principal Investigator in dialogue with the Sponsor Medical Monitor.
8. Females must not be currently pregnant or breast feeding.
9. Unlikely to comply with the study protocol.
10. Known or suspected alcohol or drug abuse within the past 6 months.
11. Received another investigational agent within 4 weeks of Day -1, or within five half-lives of Day -1, whichever is longer; or receiving any other investigational agent during this study.
12. Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol, or obscure interpretation of the trial data.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schwab, MD, Principal Investigator — Celerion; Stuart Kahn, MD, Study Director — Syntrix Biosystems
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zebala JA, Searle SL, Webster LR, Johnson MS, Schuler AD, Maeda DY, Kahn SJ. Desmetramadol Has the Safety and Analgesic Profile of Tramadol Without Its Metabolic Liabilities: Consecutive Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Trials. J Pain. 2019 Oct;20(10):1218-1235. doi: 10.1016/j.jpain.2019.04.005. Epub 2019 Apr 18. PMID 31005596

RESULTS

PARTICIPANT FLOW:
Groups:
- A-B-D-C; B-C-A-D; C-D-B-A; D-A-C-B: Treatments A, B, C and D given in the order indicated, wherein A is desmetramadol 3 x 10 mg tablets, fed; B is desmetramadol 3 x 10 mg tablets, fasted; C is desmetramadol 2 x 10 mg tablets, fasted; and D is desmetramadol 1 x 10 mg tablets, fasted. Treatments given with 240 ml water and separated by 3 days washout. Fasted treatments comprise a 10 hour fast before and 4 hours after treatment administration. Fed treatment is given 30 minutes after a standard meal.
Period: Intervention 1 (1 Day)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout 1 (3 Days)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 2 (1 Day)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout 2 (3 Days)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 3 (1 Day)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout 3 (3 Days)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 4 (1 Day)
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B
Started | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B-D-C | B-C-A-D | C-D-B-A | D-A-C-B | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 3 | 12
  Male | 4 | 2 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 2 | 5
  Not Hispanic or Latino | 5 | 5 | 5 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 1 | 5
  White | 4 | 6 | 4 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: (-/+)-M1, AUC(0-32) and AUC(Inf)
Description: The AUC(0-32) and AUC(inf) of (-/+)-M1 after each treatment (i.e., 10, 20 and 30 mg desmetramadol fasted, and 30 mg desmetramadol fed)
Time Frame: Pre-dose (0 h), and post-dose 0.5, 1.0, 1.5, 2.0, 2.5, 3.0 ,3.5, 4, 6, 8, 12, 16, 24, and 32 h.
Population: Evaluable population. The evaluable population are those subjects with calculable values for one or more of AUC0-inf (AUC0-t when appropriate) and/or Cmax.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Desmetramadol 30 mg, Fasted: While fasting a single oral dose of 30 mg desmetramadol.
  Desmetramadol: Analgesic
- Desmetramadol 30 mg, Fed: After feeding a single oral dose of 30 mg desmetramadol.
  Desmetramadol: Analgesic
Arm/Group | Desmetramadol 10 mg, Fasted | Desmetramadol 20 mg, Fasted | Desmetramadol 30 mg, Fasted | Desmetramadol 30 mg, Fed
Number analyzed (Participants) | 24 | 23 | 23 | 23
ng*hr/mL
  AUC(0-32), (-/+)-M1 | 136.0 (30.5) | 274.9 (61.3) | 408.8 (86.0) | 450.7 (103.6)
  AUC(inf), (-/+)-M1 | 138.0 (31.1) | 279.0 (62.1) | 414.6 (87.8) | 454.4 (105.4)
Statistical Analysis 1: Comparison: Desmetramadol 10 mg, Fasted vs Desmetramadol 20 mg, Fasted vs Desmetramadol 30 mg, Fasted; Analysis of dose proportionality following 10, 20 and 30 mg fasted using a mixed-effects model based on a power function: ln(dependent variable) = β1×ln(Dose) + ln(β0) + ε. Random slope and intercept. 90% CI of β1 acceptance range of 0.8-1.25 modified to account for ratio of dose levels in this study as follows: [1+ln(0.8)/ln(3), 1+ln(1.25)/ln(3)], giving acceptance range of [0.7969, 1.2031]. If the 90% CI of β1 is within [0.7969, 1.2031], dose-proportionality is proven for the PK parameter; Test type: Other; AUC(0-36) Estimate (β1) = 1.0227
Statistical Analysis 2: Comparison: Desmetramadol 10 mg, Fasted vs Desmetramadol 20 mg, Fasted vs Desmetramadol 30 mg, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; AUC(inf) Estimate (β1) = 1.0223
Statistical Analysis 3: Comparison: Desmetramadol 30 mg, Fasted vs Desmetramadol 30 mg, Fed; Analysis of food effect on desmetramadol in the evaluable population using natural logarithm-transformed PK exposure parameters of desmetramadol enantiomers following administration of 30 mg desmetramadol in the fed and fasted states; Test type: Equivalence — Absent food effect will be established if the 90% CI for the ratio of population geometric means between fed and fasted 30 mg doses, based on log-transformed data, is contained in the equivalence limits of 0.80-1.25 for AUC0-inf and Cmax; AUC(0-inf) fed/fasted ratio = 1.09, 90% CI 2-sided [1.05 to 1.12]

2. Primary Outcome: (-/+)-M1, Cmax
Description: The Cmax of (-/+)-M1 after each treatment (i.e., 10, 20 and 30 mg desmetramadol fasted, and 30 mg desmetramadol fed)
Time Frame: Pre-dose (0 h), and post-dose 0.5, 1.0, 1.5, 2.0, 2.5, 3.0 ,3.5, 4, 6, 8, 12, 16, 24, and 32 h.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Desmetramadol 10 mg, Fasted | Desmetramadol 20 mg, Fasted | Desmetramadol 30 mg, Fasted | Desmetramadol 30 mg, Fed
Number analyzed (Participants) | 24 | 23 | 23 | 23
ng/mL | 12.41 (2.59) | 24.22 (5.08) | 36.27 (7.47) | 43.42 (10.73)
Statistical Analysis 1: Comparison: Desmetramadol 10 mg, Fasted vs Desmetramadol 20 mg, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; Cmax Estimate (β1) = 0.9899
Statistical Analysis 2: Comparison: Desmetramadol 30 mg, Fasted vs Desmetramadol 30 mg, Fed; [analysis description as in outcome 1, analysis 3]; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; Cmax 90% fed/fasted ratio = 1.18, 90% CI 2-sided [1.08 to 1.28]

3. Secondary Outcome: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.
Description: Adverse events will include: 1) reports by participants; 2) observations by investigators; and 3) abnormal laboratory safety test results.
Time Frame: Participant report adverse events throughout study enrolment; investigators observe adverse events during all 11 days of inpatient treatment; laboratory safety labs are obtained on Day 11 (the final study day).
Population: Only treatment-emergent AEs (TEAEs) are summarized. A TEAE is defined as an AE that is starting or worsening at the time of or after study drug dosing. Each TEAE will be attributed to a treatment based on the onset date and time of the AE. An AE that occurs during the washout period between drugs will be considered treatment-emergent to the last drug administered prior to onset of the AE. See "Adverse Events" for data table.
Measure: Count of Participants; unit: Participants
Arm/Group | Desmetramadol 10 mg, Fasted | Desmetramadol 20 mg, Fasted | Desmetramadol 30 mg , Fasted | Desmetramadol 30 mg , Fed
Number analyzed (Participants) | 24 | 23 | 23 | 23
Participants | 3 | 4 | 5 | 6

ADVERSE EVENTS:
Time Frame: 11 days.
Arm/Group | Desmetramadol 10 mg, Fasted | Desmetramadol 20 mg, Fasted | Desmetramadol 30 mg , Fasted | Desmetramadol 30 mg , Fed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/24 | 4/23 | 5/23 | 6/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desmetramadol 10 mg, Fasted (N=24) | Desmetramadol 20 mg, Fasted (N=23) | Desmetramadol 30 mg , Fasted (N=23) | Desmetramadol 30 mg , Fed (N=23)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall retain title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the performance of the Services. Such publications shall not be made by Celerion without the prior written consent of Sponsor.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Omni-Pain-103_Protocol_v1.2 (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT04683926/Prot_SAP_000.pdf
  • Statistical Analysis Plan: SAP_F1_09Feb2021 (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04683926/SAP_001.pdf
  • Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT04683926/ICF_002.pdf